CLINICAL TRIAL: NCT01991574
Title: Study of the Effect of the Consumption of Ferric Hydroxide Adipate on Urinary Phosphorus.
Brief Title: Effect of the Consumption of Ferric Hydroxide Adipate on Urinary Phosphorus Excretion.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, dora pereira, Dr, Medical Research Council
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 6320
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Healthy; Chronic Kidney Diseases
Keywords: urinary phosphate; iron hydroxide; hypophosphatemia; phosphate binder; ferric hydroxide adipate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypophosphatemia | interventions — calcium acetate

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Methylcellulose (Placebo Comparator): On one of the study days: ingest one methylcellulose capsule with a test meal rich in phosphate.
  Interventions: Drug: Placebo
- Calcium Acetate (Active Comparator): On one of the study days: ingest 667 mg calcium acetate, equivalent to 169 mg elemental calcium, with a test meal rich in phosphate.
  Interventions: Drug: Calcium acetate
- Iron Hydroxide Adipate (Experimental): On one of the study days: ingest 800 mg ferric hydroxide adipate, equivalent to 175 mg elemental iron, with a test meal rich in phosphate.
  Interventions: Dietary Supplement: Iron Hydroxide Adipate

INTERVENTIONS:
Drug: Calcium acetate
  Arms: Calcium Acetate
Dietary Supplement: Iron Hydroxide Adipate
  Arms: Iron Hydroxide Adipate
Drug: Placebo — methylcellulose capsules
  Arms: Methylcellulose

SUMMARY:
Ferric hydroxide adipate is a ferric iron supplement containing iron hydroxide and a dietary organic acid that was developed at MRC Human Nutrition Research. We aim to determine if the ingestion of ferric hydroxide adipate with food induces a reduction in urinary phosphate concentration, compared with the administration of placebo plus the same food on a different occasion. We hypothesise that ferric hydroxide adipate binds some phosphate ions in the gastrointestinal tract, which prevents part of the phosphate load in a meal from being absorbed. On another visit, calcium will be given with the same food, as a positive control, since this element is well known to restrict dietary phosphate absorption through the formation of insoluble calcium phosphates in the gut lumen. We will compare urinary phosphate concentrations after co-ingestion of the calcium salt and food versus urinary phosphate following ferric hydroxide adipate and the same food. Additionally, the calcium data will be compared with placebo data, since a significant reduction in urinary phosphate concentrations after calcium treatment will confirm the suitability of the study design.

Finally, iron absorption from the ferric hydroxide adipate treatment will be determined by labelling this preparation with 58Fe and measuring day 14 erythrocyte 57Fe:58Fe.

The study design is: Three-way cross-over volunteer absorption study. Volunteers will not be told which treatment they receive (placebo, ferric hydroxide adipate, or supplemental calcium). Researchers co-ordinating the study on a day to day basis will be aware of treatment allocation, but analysts will not be told which samples correspond to which treatments.

ELIGIBILITY:
Inclusion Criteria:

- Males and females, aged >18 years, who are generally healthy.

Exclusion Criteria:

* Pregnancy and lactation
* iron deficiency and iron deficiency anaemia
* weight change of +/-2kg in the past month
* dysphagia
* surgery in the past three months
* cancer in the last ten years
* diabetes
* known medical and genetic conditions interfering with calcium and phosphate metabolism: e.g. hyper/hypo-parathyroidism, Fanconi syndrome, hyper/hypothyroidism (except individuals who are taking stable doses of thyroid hormones)
* chronic infection or chronic inflammation
* cardiovascular disease
* chronic respiratory disease
* abnormal renal function (based on glomerular filtration rate)
* known renal disease
* abnormal liver function/known liver disease
* hereditary haemochromatosis or haemoglobinopathies
* gastrointestinal disease
* bone disease
* hypertension
* current use of proton pump inhibitors
* use of other medication that affects mineral homeostasis (on a case by case basis, in consultation with HNR clinician)
* Extreme muscle hypertrophy (e.g. body building)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
urinary phosphate | 9 hours
  To determine if the ingestion of ferric hydroxide adipate with food induces a reduction in urinary phosphate concentration, compared with the administration of placebo plus the same food on a different occasion.

SECONDARY OUTCOMES:
iron absorption | 14 days
  iron absorption from the ferric hydroxide adipate treatment will be determined by labelling this preparation with 58Fe and measuring day 14 erythrocyte 57Fe:58Fe.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Powell, PhD, Study Chair — Medical Research Council
Locations (1):
- MRC Human Nutrition Research, Cambridge, Cambridgeshire, United Kingdom